CLINICAL TRIAL: NCT05450211
Title: Evaluation of Postoperative Analgesic Efficacy of Suprainguinal Fascia Iliaca Block Applied With Ultrasonography in Knee Arthroplasty
Brief Title: Evaluation of Postoperative Analgesic Efficacy of Suprainguinal Fascia Iliaca Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Hale Kefeli Celik, Anesthesiologist, Principal Investigator, Samsun Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: OYKU55
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Regional Anesthesia
Keywords: regional analgesia; suprainguinal fascia iliaca block; patient controlled analgesia
MeSH Terms: interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patient will not know which study group he is in. The anesthetist, who will perform the regional block, will give the block to be applied in a sealed envelope by an assistant staff outside the study, and at the same time, the patient will not know which block has been made. The anesthesiologist who made the block will not participate in the pain follow-up of the patients. Postoperative pain assessment and data collection will be performed by another investigator blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SFI (Suprainguinal fascia iliaca block) (Active Comparator): In the patient lying in the supine position, a high-frequency linear probe is inserted under sterile conditions, using an in-plane technique, 1 cm cephalad of the inguinal ligament with an 85 mm needle. Using hydro-dissection, the fascia iliaca is separated from the iliac muscle and a space is created where the needle can be advanced cranially, and the procedure will be completed by injecting local anesthetic into this space.
  When the patient whose block procedure is successful, is taken to the recovery room, controlled analgesia will be applied to the patient and he will be transferred to the ward. Tramadol HCL will be used for postoperative pain control for PCA.
  Interventions: Device: Low frequency convex probe (ESAOTE Fixed Color Doppler Ultrasonography Device, Italy); Device: Patient controlled analgesia
- Group PCA (patient controlled analgesia) (Active Comparator): No block attempt will be made to the patients in this group, and when the patient is taken to the recovery room after surgery, controlled analgesia will be administered and transferred to the ward. Tramadol HCL will be used for postoperative pain control for PCA.
  Interventions: Device: Patient controlled analgesia

INTERVENTIONS:
Device: Low frequency convex probe (ESAOTE Fixed Color Doppler Ultrasonography Device, Italy) — A low frequency convex probe (ESAOTE Fixed Color Doppler Ultrasonography Device, Italy) device will be used while blocking in group SFI.
  Arms: Group SFI (Suprainguinal fascia iliaca block)
Device: Patient controlled analgesia — Patient-controlled analgesia will be used for pain control after surgery in both groups.

SUMMARY:
It was aimed to evaluate the postoperative analgesic efficacy of the suprainguinal fascia iliaca block applied in the postoperative period in terms of 24-hour opioid consumption, pain score, additional analgesic need, and side effects and complications in the postoperative period, and to see the postoperative analgesic effectiveness of this block in patients who underwent knee arthroplasty.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is one of the major orthopedic surgeries that cause severe postoperative pain. A successful post-operative outcome is possible with strong and effective pain control followed by early mobilization and a good functional recovery.

There are many studies in the literature showing successful results regarding the effectiveness of suprainguinal fascia iliaca block on postoperative pain in pain control after hip surgery. However, there is not enough information about the use of suprainguinal fascia iliaca block in knee arthroplasty. With this study, the investigators aim to contribute to the literature on the use and effectiveness of suprainguinal fascia iliaca block in knee arthroplasty.

An identification number (ID) number will be randomly assigned to each participants, whose written consent was obtained before the surgery, when they are admitted to the postoperative recovery room. In the postoperative period, participans will be followed up with these numbers in patient follow-up. Which group the participants will be included in will be determined by the closed envelope method.

Participants who underwent unilateral knee arthroplasty will be included in the prospective and randomized study. The participants will be divided into two groups and suprainguinal fascia iliaca block and patient-controlled analgesia (Group SFI) will be applied to one group and patient-controlled analgesia (Group PCA) will be applied to the other group.

No block attempt will be made to the participants in the patient-controlled analgesia group (Group PCA), and when the patient is taken to the recovery room after surgery, patient-controlled analgesia will be administered and transferred to the ward.

Group SFI; the block procedure will be applied to the participant lying in the supine position under sterile conditions with a high-frequency linear probe (ESAOTE Fixed Color Doppler Ultrasonography Device, Italy).In the block method, 0.25% bupivacaine (Buvasin Vem İlaç, Turkey) (15 ml physiological saline + 15 ml 0.5% bupivacaine) total amount of 30 ml, same volume and same concentration will be used. The participant with the block will be followed in the recovery room and if the block is successful, PCA treatment will be started and the participant will be taken to the ward.

Evaluation of postoperative pain will be done with numerical rating scale (NRS).Pain levels will be questioned in two different ways as rest and passive moving.

ELIGIBILITY:
Inclusion Criteria: Patients,

* Having undergone unilateral knee replacement surgery under elective conditions,
* Age range of 18-75 years,
* ASA score I and II,
* Body mass index < 35kg/m²,
* written consent who agreed to participate in the study.

Exclusion Criteria: Patients,

* who do not want to be included in the study by not signing the voluntary consent form,
* Body mass index > 35 kg/m²,
* Local infection, hematoma, hernia, neoplasm etc. in the area to be blocked. found,
* Coagulopathy, hepatic or renal failure,
* Allergic to a local anesthetic agent or one of the drugs used in the study,
* Having a history of chronic opioid and corticosteroid use,
* who cannot use the patient-controlled analgesia system and have a psychiatric disease,
* with operative time less than 20 minutes and more than 120 minutes for better standardization of studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Analgesic consumption | Postoperative 24 hours
  To determine the amount of analgesic consumption in the postoperative first 24 hours with PCA in the postoperative period.

SECONDARY OUTCOMES:
Numerical Rating Scale | Postoperative 24 hours
  To determine the pain of the patients at rest and passive moving at the 1st, 3rd, 6th, 12th, 18th and 24th hours postoperatively with Numerical Rating Scale (NRS).The NRS is a segmented numerical version in which the respondent selects an integer (0-10) that best reflects the intensity of their pain. 0: no pain 1-3: mild pain 4-6: moderate pain 7-10: severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Suren, Professor, Study Chair — Samsun Research and Education Hospital
Locations (1):
- Samsun Research and Education Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Researched data and statistical analyzes will be available from the journal in which the clinical study was published.

REFERENCES:
- [Result] Seo SS, Kim OG, Seo JH, Kim DH, Kim YG, Park BY. Comparison of the Effect of Continuous Femoral Nerve Block and Adductor Canal Block after Primary Total Knee Arthroplasty. Clin Orthop Surg. 2017 Sep;9(3):303-309. doi: 10.4055/cios.2017.9.3.303. Epub 2017 Aug 4. PMID 28861197
- [Result] Desmet M, Vermeylen K, Van Herreweghe I, Carlier L, Soetens F, Lambrecht S, Croes K, Pottel H, Van de Velde M. A Longitudinal Supra-Inguinal Fascia Iliaca Compartment Block Reduces Morphine Consumption After Total Hip Arthroplasty. Reg Anesth Pain Med. 2017 May/Jun;42(3):327-333. doi: 10.1097/AAP.0000000000000543. PMID 28059869
- [Result] Hebbard P, Ivanusic J, Sha S. Ultrasound-guided supra-inguinal fascia iliaca block: a cadaveric evaluation of a novel approach. Anaesthesia. 2011 Apr;66(4):300-5. doi: 10.1111/j.1365-2044.2011.06628.x. Epub 2011 Feb 24. PMID 21401544
- [Result] Vermeylen K, Soetens F, Leunen I, Hadzic A, Van Boxtael S, Pomes J, Prats-Galino A, Van de Velde M, Neyrinck A, Sala-Blanch X. The effect of the volume of supra-inguinal injected solution on the spread of the injectate under the fascia iliaca: a preliminary study. J Anesth. 2018 Dec;32(6):908-913. doi: 10.1007/s00540-018-2558-9. Epub 2018 Sep 24. PMID 30250982